CLINICAL TRIAL: NCT04706936
Title: Novel BCMA-targeted CAR-T Cell Therapy for Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Carbiogene Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2020001474
Record Dates: First submitted 2020-12-03; First posted 2021-01-13 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: BCMA; Chimeric antigen receptor T cell; Adoptive cell therapy
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-BCMA CAR-T (CBG-002) (Experimental): All subjects were intravenous administrated with CBG-002.
  Interventions: Biological: anti-BCMA CAR-T; Drug: Cyclophosphamid; Drug: Fludarabine

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Retroviral vector-transduced autologous T cells to express anti-BCMA CAR.
  Other Names: CBG-002 CAR-T
Drug: Cyclophosphamid — 300mg/m2/d
Drug: Fludarabine — 30mg/m2/d

SUMMARY:
This study evaluates the safety and efficacy of novel BCMA-targeted CAR-T cell therapy (CBG-002) for patients with relapsed or refractory multiple myeloma (r/r MM). CBG-002 is designed based on the fourth-generation of CAR-T techonology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory multiple myeloma aged 18-75 years;
2. BCMA expression ≥50% in bone marrow samples confirmed by Flow Cytometry or IHC is positive for BCMA expression;
3. Relapsed/refractory patients who meet the following conditions:

   1. Ineffective or disease progression after receiving bortezomib (proteasome inhibitor) and lenalidomide for 3 courses;
   2. Ineffective or disease progression after receiving the original treatment plan for 3 courses;
   3. The interval between the last treatment and disease progression is more than 30 days;
   4. There is currently no indication for hematopoietic stem cell transplantation, or the patient refuses to do hematopoietic stem cell transplantation;
   5. The definition of disease progression refers to the "2014 IMWG Standards", and at least meets the following 1 items:

   e.1 Serum M protein ≥ 0.5 g/dL;

   e.2 Urine M protein ≥ 200 mg/24 h;

   e.3 If the serum FLC ratio is abnormal, the patient's FLC level ≥ 10 mg/dL (100 mg/L);

   e.4 Evaluable plasmacytoma confirmed by biopsy;

   e.5 Increase in the proportion of bone marrow plasma cells ≥25% (absolute increase ≥10%);

   e.6 Bone marrow plasma cells account for 30% of the total bone marrow cells;
4. Estimated survival time> 12 weeks;
5. The disease status can be assessed and meet at least one of the following:

   1. Serum M-protein ≥10 g/L;
   2. 24h urine M-protein ≥200mg;
   3. Serum FLC≥5mg/dL;
   4. Plasma cell tumors that can be assessed by testing or images;
   5. The proportion of bone marrow plasma cells ≥ 30%;
6. ECOG physical status score 0-1;
7. Have enough venous access for apheresis or venous blood collection, and there are no other contraindications for blood cell separation;
8. WBC ≥ 1.5×109/L; PLT ≥ 45×109/L;
9. Serum creatinine ≤ 1.5 upper limit of normal (ULN) ;
10. ALT ≤ 2.5 ULN, AST ≤ 2.5 ULN.

All laboratory test results within the above range should have no ongoing continuous supportive treatment.

Exclusion Criteria:

-

Subjects who meet any of the following criteria cannot be selected for this study:

1. Systemic treatment such as lymphatic depletion with cyclophosphamide and fludarabine within 2 weeks before enrollment or single cell collection, or cell therapy within 8 weeks before treatment;
2. HCV or HIV positive; any uncontrollable active infection, including active tuberculosis, HBV DNA level ≥1×103 copies/mL;
3. Active infections occurred within 72 hours before cleansing; as long as there is no evidence of active infection and antibiotics are not in the list of prohibited drugs, subjects who continue to use preventive antibiotics, antifungal drugs or antiviral drugs are not excluded;
4. The current systemic use of cyclosporine or steroid drugs such as dexamethasone, recent or current use of inhaled steroids is not excluded;
5. Renal insufficiency, serum creatinine>1.5 upper limit of normal (ULN);
6. Liver insufficiency, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>2.5 times ULN and direct bilirubin>1.5 times ULN;
7. Hyponatremia, blood sodium <125 mmol/L;
8. Baseline serum potassium <3.5 mmol/L (potassium supplementation can be given before participating in the study, and serum potassium recovery above this standard is not excluded);
9. Pregnant or lactating women;
10. Other serious diseases that may restrict subjects from participating in this trial (such as central nervous system disease, severe heart insufficiency, myocardial obstruction or unstable arrhythmia or unstable angina, gastric ulcer in the past 6 months , Active autoimmune diseases, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3 or 4 treatment related adverse effect | 24 weeks after last dose of CAR-T treatment
  All the CAR-T treatment related adverse events，including Dose limiting toxicity (DLT), cytokine release syndrome (CRS), CAR-T associated encephalopathy syndrome, will be assessed and graded by NCI CTCAE v 5.0.
Overall response rate (ORR) after treated by CAR-T treatment | up to 2 years after CAR-T treatment
  ORR will be assessed and graded by the international Myeloma Working Group (IMWG) Unified response criteria for multiple myeloma

SECONDARY OUTCOMES:
Pharmacokinetics of CAR-T cells (implantation endpoint) | up to 2 years after CAR-T treatment
  To assess the duration of CAR-positive T cells in circulation, the copy number of CAR DNA was measured at the preset follow-up time point. The time when the results of any two consecutive tests were negative, were recorded as the "implantation endpoint".
Overall survival | up to 2 years after CAR-T treatment
  From date of inclusion to date of progression, relapse, or death from any cause.
Progression free survival | up to 2 years after CAR-T treatment
  The length of time that a participant's disease did not progress during and after CAR-T treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741